CLINICAL TRIAL: NCT02941601
Title: A Multicenter, Phase 2 Study of Gemcitabine-Carboplatin Plus Necitumumab in Chemotherapy-Naïve Patients With Locally Advanced or Metastatic Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Gemcitabine-Carboplatin Plus Necitumumab (LY3012211) in Chemotherapy-Naïve Participants With Locally Advanced or Metastatic Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This was a strategic decision for business planning purposes and not out of concern for patient safety.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16535; I4X-MC-JFDA (Other: Eli Lilly and Company); 2016-002041-31 (EudraCT Number)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Locally Advanced Squamous Non-Small Cell Lung Cancer; Metastatic Squamous Non-Small Cell Lung Cancer
Keywords: Thoracic Neoplasms; Lung Diseases; Lung Cancer; Respiratory Tract Diseases; Respiratory Tract Neoplasms; Antineoplastic Agents; Monoclonal Antibodies
MeSH Terms: conditions — Thoracic Neoplasms; Lung Diseases; Lung Neoplasms; Respiratory Tract Diseases; Respiratory Tract Neoplasms | interventions — necitumumab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Necitumumab + Gemcitabine and Carboplatin (Experimental): Predominately European sites. Gemcitabine administered intravenously (IV) and carboplatin IV plus necitumumab IV.
  Interventions: Drug: Necitumumab; Drug: Gemcitabine; Drug: Carboplatin
- Cohort 2: Necitumumab + Gemcitabine and Carboplatin (Experimental): Predominately United States sites. Gemcitabine administered IV and carboplatin IV plus necitumumab IV.
  Interventions: Drug: Necitumumab; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Necitumumab — Administered IV
  Other Names: LY3012211
Drug: Gemcitabine — Administered IV
  Other Names: LY188011
Drug: Carboplatin — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the effectiveness and safety of gemcitabine-carboplatin plus necitumumab in chemotherapy-naïve participants with locally advanced or metastatic squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of locally advanced or metastatic NSCLC in Cohort 1 and metastatic NSCLC in Cohort 2, predominantly squamous histology. Squamous NSCLC diagnosis must be confirmed by histology or cytology local pathology report.
* Participants in Cohort 1 are required to have epidermal growth factor receptor (EGFR) protein expressing tumor (defined by local immunohistochemistry test). This is not required for participants in Cohort 2.
* Measurable disease at the time of study entry as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-1
* Have discontinued all previous treatments for cancer and recovered from the acute effects of therapy: Biologic agents (for example, antibodies) and Immunotherapy ≥4 weeks; Chest radiotherapy ≥4 weeks; Major surgery, excluding biopsy ≥4 weeks)
* The participant has archived tumor tissue available for biomarker analyses.
* Participants in Cohort 2 are required to have received 1 prior single-agent immune checkpoint inhibitor for squamous NSCLC.

Exclusion Criteria:

* The participant has nonsquamous NSCLC
* The participant has received prior anticancer therapy targeting the EGFR, vascular endothelial growth factor (VEGF), or VEGF receptor.
* The participant has received previous chemotherapy (including concurrent chemoradiation) for advanced NSCLC (participants who have received neo-adjuvant and/or adjuvant chemotherapy are eligible if the last administration occurred at least 1 year prior to start of therapy).
* The participant has brain metastases that are symptomatic or require ongoing treatment with steroids or anticonvulsants.
* The participant has a bleeding tumor.
* The participant has a history of arterial or venous thromboembolism within 3 months prior to study enrollment.
* The participant has a history or evidence of current clinically-relevant coronary artery disease of current ≥ Class III as defined by Canadian Cardiovascular Society Angina Grading Scale (Campeau 1976) or congestive heart failure of current ≥ Class III as defined by the New York Heart Association.
* The participant has experienced myocardial infarction within 6 months prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR): Percentage of Participants With a Complete or Partial Response | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Approximately 18 Months)

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline to Date of Death Due to Any Cause (Approximately 24 Months)
Progression Free Survival (PFS) | Baseline to Measured Progressive Disease or Death (Approximately 24 Months)
Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of Complete Response, Partial Response, and Stable Disease | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Approximately 24 Months)
Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab | Cycle 1 Day 1 through Cycle 6 Day 1 (Approximately 4 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- Fairview Southdale Oncology Clinic, Edina, Minnesota, United States
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haine-St.- Paul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roeselare
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bamberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avellino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Messina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bebington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

IPD SHARING:
Plan to Share IPD: No